CLINICAL TRIAL: NCT03633500
Title: Effectiveness of Mother's Own Colostrum and Breast Milk as Oral Immunotherapy and on the Feeding Behaviors and Clinical Outcome Among Preterm Infants
Brief Title: Effectiveness of Oral Immunotherapy Among Preterm Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Adan Hospital Kuwait (Industry)
Responsible Party: Principal Investigator, Shiney Easo, Staff Nurse,, Al Adan Hospital Kuwait
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 545/2017
Record Dates: First submitted 2018-05-31; First posted 2018-08-16 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Feeding Behavior; Late-Onset Neonatal Sepsis
Keywords: Colostrum; Oral immune therapy; Preterm; Oral feeding; Sepsis
MeSH Terms: conditions — Feeding Behavior; Neonatal Sepsis; Premature Birth; Sepsis

STUDY DESIGN:
Intervention Model Description: the intervention is carried out among preterm babies below 33 weeks of gestation or weight less than 1500gm
Who Masked: Care Provider, Investigator
Masking Description: Block size and number of blocks: the sample size estimated for the study was 48 the size of the blocks is fixed in nature. Hence there are 6 blocks with a block size of 8 preterm babies each in every block.
  Allocation ratio: one to one allocation ratio will be used for the study. Since the block size is 8 and one to one allocation was used, each block consist of 4 babies in each group (experimental:4, control =4) Sequence generation: 6 sets of random sequence will be generated with the help of research randomizer, an online random number generator. The sequence will be generated by an external member, who was not directly involved in the study.
  Allocation concealment: Concealed allocation was achieved using sequentially Numbered, Opaque, Sealed Envelopes (SNOSESs). SNOSESs were prepared by an external member, who was not a part of study and kept in an opaque envelope.
  Blinding: is done by covering the syringe with adhesive silk tape.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterile water (Placebo Comparator): Sterile water: Started by six hours of age, In the control arm, 0.2 ml of sterile water is instilled into the posterior buccal cavity in aliquots of 0.1 ml over a 30 second period. The liquid is given time to get absorbed, any pooled liquid is swabbed in the infants' cheek and gum. This is performed every 4 hours until independent safe cup feeds, breastfeed or bottle feed is established consistently for 48 hours.
  Interventions: Other: Sterile water
- Breastmilk (Experimental): Breastmilk. This is started at 6 hours of age at the earliest; breast milk: 0.2 ml of mothers' own colostrum/ breast milk is instilled into the posterior buccal cavity in aliquots of 0.1 ml over a 30 second period. The colostrum is given time to get absorbed, any pooled milk is swabbed in the infants' cheek and gum. This is performed every 4 hours until independent safe cup feeds, breastfeed or bottle feed is established consistently for 48 hours.
  Interventions: Biological: Breastmilk

INTERVENTIONS:
Other: Sterile water — Placebo Comparator: Sterile water: 0.2 ml of sterile water is instilled into the posterior buccal cavity in aliquots of 0.1 ml over a 30 second period. The liquid is given time to get absorbed, any pooled liquid is swabbed in the infants' cheek and gum. This is performed every 4 hours until independent safe cup feeds, breastfeed or bottle feed is established consistently for 48 hours.
  Other Names: Placebo
  Arms: Sterile water
Biological: Breastmilk — Experimental: Breastmilk: 0.2 ml of mothers' own colostrum/ breast milk is instilled into the posterior buccal cavity in aliquots of 0.1 ml over a 30 second period. The colostrum is given time to get absorbed, any pooled milk is swabbed in the infants' cheek and gum. This is performed every 4 hours until independent safe cup feeds, breastfeed or bottle feed is established consistently for 48 hours. independently sucks at breast, bottle or cup feed
  Other Names: experimental
  Arms: Breastmilk

SUMMARY:
The aim of the study is to assess the effectiveness of OIT with colostrum on the feeding behavior and Clinical Outcome of Late-onset sepsis and Necrotizing enterocolitis

DETAILED DESCRIPTION:
A randomized placebo-controlled double-blinded study in preterm infants < 32+6 weeks' gestation or Birth weight < 1500 g who are admitted to NICU.

Exclusion criteria include infants with congenital anomalies, out born infants, infants of single mothers with unknown partners (mother is separated from preterm infants based on the state law) and infants admitted beyond 48 hours of age, confirmed immunodeficiency disorder, Inborn Error of Metabolism, parental refusal to participate. The infants who have overt bleeding, thrombocytopenia < 50,000/mm3 or are critically ill requiring multiple inotropes in high doses, on High frequency ventilation and inhaled nitric oxide and infants with congenital surgical abdomen are excluded from the study.

An informed parental consent is obtained at the initial post-natal visit. Each neonate is then randomly assigned to the placebo or intervention group per the block randomization generated using a computer-generated allocation sequence. Allocation is concealed from all involved investigators, bedside nurses, doctors, parents and outcome assessors except the International Board Certified Lactation Consultant (IBCLC) assigned to allocate the intervention. The IBCLC is not an investigator in the study.

Intervention group:

Colostrum that is fresh or refrigerated is collected by the IBCLC and prepared using 1cc syringes which are labeled with patient identification data, date and time of milk expression. These syringes are concealed using adhesive silk tapes and handed over to the bedside nurse. The tip of the syringe is placed towards the posterior end of the buccal cavity, colostrum/breastmilk is slowly squirted in aliquots of 0.1 ml of the milk into the area . This is to be done slowly drop by drop over a 30 s period. The milk should not pool in the buccal cavity. If it pools, give a few seconds to get absorbed and the rest may be manually rubbed using a swab along the gums and the inner surface of the buccal cavity for 10 seconds with two strokes in each area. Repeat the procedure on the opposite side. If the colostrum was refrigerated the syringe may be kept in the warm incubator for five minutes before administering.

OIT will be initiated as soon after birth as colostrum is available no earlier than six hours of age and continued every 4 hours as available. OIT may be provided in babies who are kept nil per oral and is to be continued even when enteral feeding has been ordered to get a minimum of 20 doses and can be continued until the baby reaches full oral feeding.

Control group: The control group will receive 0.2 ml of sterile water that will be prepared and applied in an identical manner and frequency to that among the intervention group. This will be started at six hours of age to avoid disclosure of intervention and control group. However, as soon as Mother's milk is available it will be initiated enterally.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies below 33 weeks (32+6) weeks of gestation
* Birth weight <1500 g

Exclusion Criteria:

* Preterm babies with congenital anomalies
* Preterm babies with congenital infection like pneumonia.
* Babies born in other hospitals
* Babies of single mothers with unknown partners
* Confirmed immunodeficiency disorder,
* Inborn Error of Metabolism,
* Parental refusal to participate.
* Preterm babies who have overt bleeding

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Feeding Behaviors | Birth to 45 weeks post menstrual age
  feeding behaviour is assessed using a questionaire on feeding behaviour. it consist of feed interruptions due to intolerance, time to reach full enteral feeding, time to independent oral feeds via direct breastfeed, cup or syringe feed or bottle feed consistently for 48 hours safely.

SECONDARY OUTCOMES:
Late onset sepsis | Birth to 45 weeks post menstrual age
  late onset sepsis is measured using questionnaire on clinical outcome . it consist of culture proven sepsis and number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Shiney Easo, masters, Principal Investigator — AL Adan Hospital
Locations (1):
- Shiney Easo, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No